CLINICAL TRIAL: NCT05880069
Title: Clinical Outcomes in Patients With Infection by Resistant Microorganism
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hospital Universitario Virgen Macarena (Other)
Collaborators: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: PRIMAVERA
Record Dates: First submitted 2023-05-04; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Pneumonia; Bloodstream Infection; Urinary Tract Infections; Skin Infection; Surgical Site Infection; Staphylococcus Aureus; Klebsiella Pneumonia; Escherichia Coli; Enterococcus Faecium Infection; Acinetobacter Infections; Pseudomonas Aeruginosa
MeSH Terms: conditions — Pneumonia; Sepsis; Urinary Tract Infections; Cellulitis; Surgical Wound Infection; Staphylococcal Infections; Escherichia coli Infections; Acinetobacter Infections; Pseudomonas Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Drug-resistant pathogen: Individuals of all ages with the target pathogen, resistance phenotype, and infection site combinations as follows:
  1. P. aeruginosa, carbapenems resistant: BSI
  2. A. baumannii, carbapenems resistant: BSI
  3. E. coli, 3rd generation cephalosporins resistant: BSI and UTI
  4. K. pneumoniae, 3rd generation cephalosporins resistant: BSI
  5. K. pneumoniae, carbapenems resistant: BSI
  6. S. aureus, methicillin resistant: BSI, pneumonia, SSI and SSTI
  7. E faecium, vancomycin resistant: BSI
  8. Enterobacterales, 3rd generation cephalosporins resistant: BSI
  Interventions: Other: Pathogen resistant phenotype
- Drug-susceptible pathogen: Individuals of all ages with the target pathogen, susceptible phenotype, and infection site combinations as follows:
  1. P. aeruginosa, carbapenems susceptible: BSI
  2. A. baumannii, carbapenems susceptible: BSI
  3. E. coli, 3rd generation cephalosporins susceptible: BSI and UTI
  4. K. pneumoniae, 3rd generation cephalosporins susceptible: BSI
  5. K. pneumoniae, carbapenems susceptible: BSI
  6. S. aureus, methicillin susceptible: BSI, pneumonia, SSI and SSTI
  7. E faecium, vancomycin susceptible: BSI
  8. Enterobacterales, 3rd generation cephalosporins susceptible: BSI
  Interventions: Other: Pathogen resistant phenotype
- No infection: Individuals of all ages without the infection under study

INTERVENTIONS:
Other: Pathogen resistant phenotype — Drug resistant phenotype of the target pathogen under study
  Groups: Drug-resistant pathogen; Drug-susceptible pathogen

SUMMARY:
The goal of this individual patient data meta-analysis is to estimate the attributed and the associated health burden related to bloodstream infections, pneumonia, skin and soft tissue infections, surgical site infections and urinary tract infections, caused by target drug-resistant pathogens, in high income countries.

The main question[s] it aims to answer are:

* Are common infections caused by drug-resistant pathogens associated with an increased health burden, when compared with individuals with the same infection caused by a susceptible strain (attributed burden)?
* Are common infections caused by drug-resistant pathogens associated with an increase health burden, when compared with individuals without the infection under study (associated burden)?

ELIGIBILITY:
Inclusion Criteria:

* Individuals of all ages
* Individuals with hospital acquired, community acquired, or healthcare associated infections
* Individuals treated at hospital level, community, or long-term care facilities
* Individuals with the targeted pathogen, resistance phenotype, and infection site combinations under study

Exclusion Criteria:

* Individuals with infections in the following systems: central nervous system, genital system, pelvic infections and head and neck infections
* Individuals with the following specific primary infections: endocarditis, upper respiratory tract infections, lung abscess
* Individuals with bacterial infections not included in the table of pathogens of interest, polymicrobial infections except for intraabdominal infections, fungal infections, parasitic infections, viral infections, mycobacterial infections, sexually transmitted diseases, and zoonotic infections

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 1. Individuals of all ages with the target pathogen, resistance phenotype, and infection site combinations as follows:
     * P. aeruginosa, carbapenems resistant: BSI
     * A. baumannii, carbapenems resistant: BSI
     * E. coli, 3rd generation cephalosporins resistant: BSI and UTI
     * K. pneumoniae, 3rd generation cephalosporins resistant: BSI
     * K. pneumoniae, carbapenems resistant: BSI
     * S. aureus, methicillin resistant: BSI, pneumonia, SSI and SSTI
     * E faecium, vancomycin resistant: BSI
     * Enterobacterales, 3rd generation cephalosporins resistant: BSI
  2. Individuals of all ages with the same infection caused by the target drug-susceptible pathogen
  3. Individuals of all ages without the infection under study
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Mortality | Through study completion, an average of 1 year
  Death any time after infection, during the follow-up time of the original study.

SECONDARY OUTCOMES:
Number of participants with ICU admission | Through study completion, an average of 1 year
  Need for an admission in ICU setting for more than 24 hours after infection onset.
Number of participants with clinical cure | Through study completion, an average of 1 year
  Absence of symptoms after completion of an antibiotic treatment course.
Number of participants with microbiological cure | Through study completion, an average of 1 year
  No isolation of the causal microorganisms after completion of an antibiotic treatment course.
Number of participants with recurrence of infection | Through study completion, an average of 1 year
  Infection with the same organism after more than two weeks of the initial infection.
Number of participants with superinfection | Through study completion, an average of 1 year
  Other infections different from the one under assessment.
Number of participants with cognitive impairment / disability | Through study completion, an average of 1 year
  Impairment is any temporal or permanent loss of function; disability is a restriction or inability to perform a normal activity resulting from an impairment. Assessed using Center for Epidemiologic Studies Depression Scale (CES-D), Mini-Mental State Examination (MMSE) or Trail Making Test (TMT).

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Rodríguez-Baño, MD PhD, Study Director — Unidad Clínica de Enfermedades Infecciosas, Microbiología. Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided